CLINICAL TRIAL: NCT01593852
Title: X-ray Dose Reduction in Electrophysiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL39479.060.012
Record Dates: First submitted 2012-03-27; First posted 2012-05-08 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Arrhythmias, Cardiac
Keywords: X-rays; Cardiac Electrophysiology; Image Processing, Computer-Assisted; Catheter Ablation
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular X-ray dose settings (Active Comparator): For patients in this group x-ray images are acquired with regular dose settings of the x-ray system and regular image processing
  Interventions: Radiation: Regular image processing
- Reduced X-ray dose settings (Experimental): For patients in this group x-ray images are acquired with reduced dose settings of the x-ray system and advanced image processing
  Interventions: Radiation: Advanced image processing

INTERVENTIONS:
Radiation: Advanced image processing — Acquisition of x-ray images with reduced X-ray dose and advanced image processing
  Arms: Reduced X-ray dose settings
Radiation: Regular image processing — Acquisition of x-ray images with regular X-ray dose and regular image processing
  Arms: Regular X-ray dose settings

SUMMARY:
Allura Clarity is a novel X-ray imaging technology, that combines advanced real-time image noise reduction algorithms, with state-of-the-art hardware to reduce patient entrance dose significantly. This is realized by anatomy-specific optimization of the full acquisition chain (grid switch, beam filtering, pulse width, spot size, detector and image processing engine) for every clinical task individually. Furthermore, smaller focal spot sizes and shorter pulses are used, which are known to positively influence image quality .

The primary aim of this study is to verify if a significant reduction in total procedural X-ray dose during electrophysiological interventions can be achieved by using advanced image processing (Allura Clarity).

DETAILED DESCRIPTION:
X-ray dose and image quality are related by laws of physics. Low dose and high image quality cannot be achieved at the same time. However, image processing algorithms can help an x-ray system to acquire images with lower dose without influencing image quality or achieving higher image quality with equal dose.

In order to introduce a dose reduction technology the most important aspect is to validate the diagnostic image information. Philips has developed a new algorithm that is capable to process images with similar image quality but acquired at lower dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart rhythm disturbances undergoing an interventional treatment for their heart rhythm disturbance
* Patients who are allowed, able, willing to and have provided informed consent
* Patients to be treated with ablation for atrial fibrillation (paroxysmal, persistent or permanent), atypical atrial flutter or patients to be treated with ablation for ischemic or non-ischemic ventricular tachycardia
* Patients who are treated in heart catheterization room 5 (HCK5) of the Catherina Hospital

Exclusion Criteria:

* Patients under 18 years of age.
* Patient who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Dekker, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis, Eindhoven, Netherlands

REFERENCES:
- [Result] Dekker LR, van der Voort PH, Simmers TA, Verbeek XA, Bullens RW, Veer MV, Brands PJ, Meijer A. New image processing and noise reduction technology allows reduction of radiation exposure in complex electrophysiologic interventions while maintaining optimal image quality: a randomized clinical trial. Heart Rhythm. 2013 Nov;10(11):1678-82. doi: 10.1016/j.hrthm.2013.08.018. Epub 2013 Aug 22. PMID 23973946

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced X-ray Dose Settings: For patients in this group x-ray images are acquired with reduced dose settings of the x-ray system and advanced image processing
  Advanced image processing : Acquisition of x-ray images with reduced X-ray dose and advanced image processing
Period: Overall Study
Arm/Group | Reduced X-ray Dose Settings | Regular X-ray Dose Settings
Started | 68 | 68
Completed | 68 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced X-ray Dose Settings | Regular X-ray Dose Settings | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (14) | 65 (9) | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 50 | 51 | 101
Region of Enrollment [Number; unit: participants]
  Netherlands | 68 | 68 | 136

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Dose Area Product (DAP) Value
Description: Percentage reduction of reduced X-ray dose settings (Allura Clarity) vs. regular X-ray dose settings (AlluraXper) in DAP.
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: Gy*cm^2
Groups:
- Reduced X-ray Dose Settings (Allura Clarity): For patients in this group x-ray images are acquired with reduced dose settings of the x-ray system and advanced image processing
  Advanced image processing : Acquisition of x-ray images with reduced X-ray dose and advanced image processing
- Regular X-ray Dose Settings (AlluraXper): For patients in this group x-ray images are acquired with regular dose settings of the x-ray system and regular image processing
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Number analyzed (Participants) | 68 | 68
Gy*cm^2 | 8.8 [4.62 to 12.80] | 15.3 [9.14 to 25.53]
Statistical Analysis 1: Comparison: Reduced X-ray Dose Settings (Allura Clarity) vs Regular X-ray Dose Settings (AlluraXper); Test type: Non-Inferiority or Equivalence — Based on historical dose observations, a sample size of 68 patients per study group (i.e. 62 evaluable patients for 10% dropout rate) for a total of 136 patient randomized will allow for 80% power to detect for approximately 40% reduction in dose area product (DAP). This sample size will allow for detection of approximately 40% reduction in air kerma (AK). No adjustment for multiple endpoints was performed as both endpoints are assessing radiation dose; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Staff Dose Measured by DoseAware and Electronic Personal Dosimeter (EPD)
Description: Staff dose measured by Electronic Personal Dosimeter (EPD) worn by the operator over the lead apron (EPD operator) and the other mounted at a fixed location in the EP laboratory (EPD fixed)
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: µSv
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Number analyzed (Participants) | 68 | 68
µSv
  EPD operator | 3 [1.0 to 6.3] | 6 [3.3 to 10.0]
  EPD fixed | 10 [5.8 to 18.0] | 19 [9.0 to 38.5]

3. Secondary Outcome: Physician Professional Judgment on Procedural Success
Description: Measurement of professional judgment (yes/no) of the treating physician.
Time Frame: Day 0
Measure: Number; unit: percentage of procedural success
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Number analyzed (Participants) | 68 | 68
percentage of procedural success | 91 | 91

4. Secondary Outcome: Procedure Duration
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Number analyzed (Participants) | 68 | 68
minutes | 160 (58) | 162 (58)

5. Secondary Outcome: Fluoroscopy Time
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Number analyzed (Participants) | 68 | 68
minutes | 24 (13) | 26 (13)

6. Secondary Outcome: Physician Professional Judgment on Adequacy of Images for Performing the EP Procedure
Description: If fluoroscopy time (see results in other secondary outcomes), number of exposure frames (see below) and procedure duration (see results in other secondary outcomes) are equivalent between the two groups, this will indicate that image quality (IQ) is equally adequate in both groups.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: Number of exposure frames
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Number analyzed (Participants) | 68 | 68
Number of exposure frames | 83 (89) | 61 (66)

7. Secondary Outcome: Usage of Physician Controlled Dose Settings
Description: In both groups, default fluoroscopy dose settings were 'low', but could be changed by the operator to a medium or high setting for better imaging. The necessity to increase fluoroscopy dose for better imaging to medium or high was registered as a percentage of total number of fluoroscopy frames.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: percentage of total # of fluoro frames
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Number analyzed (Participants) | 68 | 68
percentage of total # of fluoro frames
  Low | 86 (28) | 88 (20)
  Medium | 2 (8) | 2 (9)
  High | 12 (24) | 9 (19)

8. Secondary Outcome: Serious Adverse Events
Time Frame: Day 0 if any
Measure: Number; unit: participants
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Number analyzed (Participants) | 68 | 68
participants | 1 | 0

9. Primary Outcome: Cumulative Air Kerma (AK) Value
Description: Percentage reduction of reducted X-ray dose settings (Allura Clarity) vs. regular X-ray dose settings (AlluraXper) in AK.
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: mGy
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Number analyzed (Participants) | 68 | 68
mGy | 75 [42.85 to 122.73] | 126 [85.79 to 226.40]
Statistical Analysis 1: Comparison: Reduced X-ray Dose Settings (Allura Clarity) vs Regular X-ray Dose Settings (AlluraXper); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During procedure
Arm/Group | Reduced X-ray Dose Settings (Allura Clarity) | Regular X-ray Dose Settings (AlluraXper)
Serious Adverse Events (participants affected / at risk) | 1/68 | 0/68
Other Adverse Events (participants affected / at risk) | 0/68 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced X-ray Dose Settings (Allura Clarity) (N=68) | Regular X-ray Dose Settings (AlluraXper) (N=68)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No